CLINICAL TRIAL: NCT03729921
Title: Comparison of Efficacy and Safety of Gastric Variceal Ligation Versus Gastric Variceal Obturation for Secondary Prophylaxis of Gastric Varices
Brief Title: Gastric Variceal Ligation Versus Gastric Variceal Obturation for Secondary Prophylaxis of Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSY-GVL&GVO
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Gastroesophageal Varices; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gastric variceal obturation (Active Comparator): gastric variceal obturation
  Interventions: Procedure: gastric variceal obturation
- gastric variceal ligation (Experimental): gastric variceal ligation
  Interventions: Procedure: gastric variceal ligation

INTERVENTIONS:
Procedure: gastric variceal ligation — The highest point of the variceal vein was used as the primary ligation site. If the input vein was not obvious, the edge of the variceal vein was ligated. The variceal veins were ligated with a 6-ring ligation device, and more than 18 rings rubber bands could be applied in one session. GVL was performed regularly until varices were obliterated or reduced to residual small varices, which could not be ligated. The residual small varices was treated by cyanoacrylate injection.
  Arms: gastric variceal ligation
Procedure: gastric variceal obturation — Gastric varices were uniformly treated via the sandwich technique, which starts with an injection of lauromacrogol, followed by N-butyl cyanoacrylate, then finished with flush of lauromacrogol. The number of injection sites and volume of lauromacrogol and cyanoacrylate used, directly correlated with the size of the varix. Multiple injection sites were chosen in attempt to obliterate the varix or varices in one session. Volume of lauromacrogol used ranged from 2-10ml, while that of cyanoacrylate ranged from 0.5-2ml, per injection site.
  Arms: gastric variceal obturation

SUMMARY:
The investigators establish a randomized controlled clinical trial, comparing the efficacy and prognosis of GVL and GVO in secondary prevention of GVs, especially in patients with portosystemic shunting, and exploring the endoscopic treatment selection of different types of GVs.

Outcome expectations: Compared with glue injection, endoscopic ligation for secondary prevention of gastric varices is safe and effective, especially in patients with portosystemic shunting.

DETAILED DESCRIPTION:
Gastric varices (GVs) is a common complication of portal hypertension, with an incidence of 20%. Though the bleeding rate of GVs (25%) is lower than that of Esophageal varices (EVs), the mortality rate is higher due to greater GVs rupture and less space for endoscopic intervention. In addition, in 30% of patients with GVs, the possibility of treatment failure exists.

Guidelines differ on endoscopic treatment for secondary prevention of GVs.Current studies suggest that EVL, due to its low incidence of complications, is suitable for GOV1, while it is still controversial for the treatment of gastric varices. Compared with glue, the advantage of ligation is that it can avoid serious complications caused by glue injection, such as ectopic embolization, large ulcer and sepsis. As there are few studies comparing GVL and GVO in secondary prevention of gastric varices, the treatment methods are different, and the treatment effect is controversial. In addition, the choice of treatment for different types of GVs needs further study.

The investigators establish a randomized controlled clinical trial, comparing the efficacy and prognosis of GVL and GVO in secondary prevention of GVs, especially in patients with portosystemic shunting, and exploring the endoscopic treatment selection of different types of GVs.

Outcome expectations: Compared with glue injection, endoscopic ligation for secondary prevention of gastric varices is safe and effective, especially in patients with portosystemic shunting.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age；Past history of gastroesophageal variceal hemorrhage confirmed by an endoscopic examination

Exclusion Criteria:

* Patients who are not suitable for endoscopic treatment judged by the clinician; Patients who are not suitable for the ligation treatment because of scar change by repeated glue injection; Patients with acute hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Rate of rebleeding | 6 months
  New onset of hematemesis, coffee-ground vomitus, hematochezia,or melena,with an increasing pulse rate over 100 beats/min and decreasing blood pressure below 90 mmHg after a 24-hour period of stable vital signs and hemoglobin after endoscopic treatment.

SECONDARY OUTCOMES:
Rate of GV eradication | 6 months
  non-visualization of patent GV
Incidence of complications | 6 months
  Huge ulcer on GV, spontaneous bacterial peritonitis, bacteremia
mortality | 6 months
  Survival situation of patience